CLINICAL TRIAL: NCT03631784
Title: A Phase 2 Trial of Pembrolizumab (MK-3475) in Combination With Platinum Doublet Chemotherapy and Radiotherapy for Participants With Unresectable, Locally Advanced Stage III Non-Small Cell Lung Cancer (NSCLC) (KEYNOTE-799)
Brief Title: A Trial of Pembrolizumab in Combination With Chemotherapy and Radiotherapy in Stage III NSCLC (KEYNOTE-799, MK-3475-799)
Acronym: KEYNOTE-799
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3475-799; MK-3475-799 (Other: MSD Protocol Number); 2018-000714-37 (EudraCT Number)
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Results first posted 2022-11-02 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1 (PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Paclitaxel; Cisplatin; Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): Participants received 1 cycle of carboplatin area under the curve (AUC) 6 mg/mL/min with paclitaxel 200 mg/m^2 and pembrolizumab 200 mg on Day 1. Approximately 3 weeks later, participants received carboplatin AUC 2 mg/mL/min with paclitaxel 45 mg/ m^2 administered weekly for 6 weeks along with 2 cycles of pembrolizumab 200 mg administered every 3 weeks (Q3W) in conjunction with standard thoracic radiotherapy (TRT) (60 Gray [Gy] in 2 Gy fractions administered 5 days per week for 6 weeks). Participants then received 14 additional cycles of pembrolizumab 200 mg administered Q3W. 1 cycle=21 days.
  Interventions: Drug: Pembrolizumab 200 mg; Drug: Paclitaxel 45 mg/m^2; Drug: Carboplatin AUC6; Radiation: Thoracic Radiation Therapy (TRT); Drug: Paclitaxel 200 mg/m^2; Drug: Carboplatin AUC2
- Cohort B (Experimental): Participants received 3 cycles of cisplatin 75 mg/m^2 with pemetrexed 500 mg/m^2 and pembrolizumab 200 mg on Day 1 of each cycle. Treatment was given in conjunction with standard TRT (60 Gy in 2 Gy fractions administered 5 days per week for 6 weeks) in cycles 2 and 3. Participants then received 14 additional cycles of pembrolizumab 200 mg administered Q3W. 1 cycle=21 days.
  Interventions: Drug: Pembrolizumab 200 mg; Drug: Cisplatin 75 mg/m^2; Drug: Pemetrexed 500 mg/m^2; Radiation: Thoracic Radiation Therapy (TRT)

INTERVENTIONS:
Drug: Pembrolizumab 200 mg — Pembrolizumab 200 mg intravenous (IV) infusion on Days 1 of each 3-week cycle for up to 17 cycles
  Other Names: MK-3475
Drug: Paclitaxel 45 mg/m^2 — Paclitaxel 45 mg/m^2 IV infusion on Days 1, 8, 15 of each 3-week cycle for Cycles 2, and 3 during radiation therapy.
  Arms: Cohort A
Drug: Carboplatin AUC6 — Carboplatin AUC6 IV infusion on Day 1 of the 21-day cycle for Cycle 1.
  Arms: Cohort A
Drug: Cisplatin 75 mg/m^2 — Cisplatin 75 mg/m^2 IV infusion on Day 1 of each 21-day cycle for Cycles 1, 2, 3.
  Arms: Cohort B
Drug: Pemetrexed 500 mg/m^2 — Pemetrexed 500 mg/m^2 IV infusion on Day 1 of each 21-day cycle for Cycles 1, 2, and 3.
  Arms: Cohort B
Radiation: Thoracic Radiation Therapy (TRT) — The target total dose of TRT will be 60 Gy in 30 daily fractions of 2 Gy, prescribed to the planning target volume.
Drug: Paclitaxel 200 mg/m^2 — Paclitaxel 200 mg/m^2 IV infusion on Day 1 of the 21-day cycle of Cycle 1.
  Arms: Cohort A
Drug: Carboplatin AUC2 — Carboplatin AUC2 IV infusion on Day 1, 8, 15 for Cycles 2 and 3 during radiation therapy.
  Arms: Cohort A

SUMMARY:
This is a trial in adult participants with unresectable, locally advanced, Stage III non-small cell lung cancer (NSCLC) treated with pembrolizumab in combination with platinum doublet chemotherapy and standard thoracic radiotherapy followed by pembrolizumab monotherapy. The primary hypothesis of the trial is that within each platinum doublet chemotherapy cohort, the percentage of participants who develop Grade 3 or higher pneumonitis is ≤10% and estimation of objective response rate (ORR) by blinded independent central review (BICR).

ELIGIBILITY:
Inclusion Criteria:

* Male/female participants, who are at least 18 years of age on the day of signing informed consent with previously untreated, unresectable, pathologically confirmed NSCLC and Stage IIIA, IIIB or IIIC NSCLC by American Joint Committee on Cancer Version 8.
* No evidence of metastatic disease by whole body positron emission tomography/computed tomography (PET/ CT) scan, diagnostic quality CT scan, and brain imaging.
* Have measurable disease per RECIST 1.1 as assessed by the local site investigator/radiology.
* Have provided tumor tissue sample (core, incisional, or excisional biopsy).
* Have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Have adequate pulmonary function test (PFT)
* Have adequate organ function
* A male participant must agree to use contraception through the end of treatment and refrain from donating sperm during this period.
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and if participant is a woman of childbearing potential (WOCBP), agrees to follow the contraceptive guidance as provided in the protocol through the end of treatment.

Exclusion Criteria:

* A WOCBP who has a positive urine pregnancy test within 72 hours prior to treatment allocation
* Has small cell lung cancer.
* Has had documented weight loss >10% in the preceding 3 months.
* Participants whose radiation treatment plans are likely to encompass a volume of whole lung receiving >20 Gy in total (V20) of more than 31% of lung volume.
* Has received prior radiotherapy to the thorax, including radiotherapy to the esophagus or for breast cancer.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent (programmed cell death protein 1 [PD-1] and its ligands, programmed cell death ligand 1 (PD-L1) and programmed cell death ligand 2 [PD-L2]) or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).
* Has received a live vaccine within 30 days prior to the first dose of study drug.
* Has had an allogenic tissue/solid organ transplant.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg prednisone daily or equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study drug.
* Has a known additional malignancy that is progressing or has required active treatment within the past 5 years.
* Has severe hypersensitivity (Grade 3 or higher) to pembrolizumab and/or any of its excipients.
* Has a known severe hypersensitivity (Grade 3 or higher) to any of the study chemotherapy agents and/or to any of their excipients.
* Has an active autoimmune disease that has required systemic treatment in past 2 years (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs).
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease that requires steroids.
* Has an active infection requiring systemic therapy.
* Has a known history of human immunodeficiency virus (HIV) infection. HIV testing is not required unless mandated by local health authority.
* Has a known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.
* Has a known history of active tuberculosis (TB; Bacillus tuberculosis).
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Has a known psychiatric or substance abuse disorder that would interfere with cooperating with the requirements of the study.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study through the end of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2021-10-18 (Actual); Study Completion 2024-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (56):
- United States (10):
  - St Joseph Heritage Healthcare ( Site 1403), Santa Rosa, California
  - North Shore University Health System ( Site 1413), Evanston, Illinois
  - Parkview Cancer Institute ( Site 1415), Fort Wayne, Indiana
  - UMass Memorial Medical Center ( Site 1417), Worcester, Massachusetts
  - Henry Ford Hospital ( Site 1418), Detroit, Michigan
  - St. Francis Cancer Treatment Center ( Site 1421), Grand Island, Nebraska
  - Rutgers Cancer Institute of New Jersey ( Site 1422), New Brunswick, New Jersey
  - CTCA Southwestern ( Site 1428), Tulsa, Oklahoma
  - Fox Chase Cancer Center ( Site 1433), Philadelphia, Pennsylvania
  - Sanford Cancer Center Oncology Clinic ( Site 1434), Sioux Falls, South Dakota
- Australia (4):
  - Blacktown Hospital Western Sydney Local Health District ( Site 0204), Blacktown, New South Wales
  - MNCCI Port Macquarie Base Hospital ( Site 0200), Port Macquarie, New South Wales
  - Southern Medical Day Care Centre ( Site 0201), Wollongong, New South Wales
  - Ballarat Health Services ( Site 0206), Ballarat, Victoria
- France (9):
  - C.H. de Saint Quentin ( Site 0306), Saint-Quentin, Aisne
  - Clinique Clairval ( Site 0311), Marseille, Bouches-du-Rhone
  - CHU Jean Minjoz ( Site 0301), Besançon, Doubs
  - Institut du Cancer de Montpellier ( Site 0300), Montpellier, Herault
  - C.H.R.U. de Rennes. Hopital de Pontchaillou ( Site 0302), Rennes, Ille-et-Vilaine
  - ICO Centre Paul Papin ( Site 0309), Angers, Maine-et-Loire
  - Centre Jean Perrin ( Site 0304), Clermont-Ferrand, Puy-de-Dome
  - Clinique de L'Europe ( Site 0308), Amiens, Somme
  - Institut de Cancerologie Gustave Roussy ( Site 0305), Villejuif, Val-de-Marne
- Germany (8):
  - Thoraxklinik Heidelberg gGmbH am Universitaetsklinikum Heidelberg ( Site 0404), Heidelberg, Baden-Wurttemberg
  - Universitatsklinikum Mannheim GmbH ( Site 0413), Mannheim, Baden-Wurttemberg
  - Augusta-Kranken-Anstalt Bochum ( Site 0401), Bochum, North Rhine-Westphalia
  - Bethanien Krankenhaus Moers ( Site 0406), Moers, North Rhine-Westphalia
  - Klinikum Chemnitz gGmbH ( Site 0410), Chemnitz, Saxony
  - LungenClinic Grosshansdorf GmbH ( Site 0408), Großhansdorf, Schleswig-Holstein
  - Charite Universitaetsmedizin Berlin - Campus-Virchow-Klinikum ( Site 0414), Berlin
  - Katholisches Marienkrankenhaus gGmbH ( Site 0411), Hamburg
- Auckland City Hospital ( Site 0700), Auckland, New Zealand
- Poland (5):
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka ( Site 0811), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Osrodek Badan Klinicznych przy Szpitalu Specjalistycznym ( Site 0802), Krakow, Lesser Poland Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie ( Site 0800), Warsaw, Masovian Voivodeship
  - Szpital Morski im. PCK. Szpitale Pomorskie Sp. Z o.o ( Site 0812), Gdynia, Pomeranian Voivodeship
  - Szpital Wojewodzki w Koszalinie im. Mikolaja Kopernika ( Site 0813), Koszalin, West Pomeranian Voivodeship
- Russia (4):
  - Republican Clinical Oncology Dispensary of Republic of Bashkortostan ( Site 0903), Ufa, Baskortostan, Respublika
  - Blokhin National Medical Oncology ( Site 0902), Moscow, Moscow
  - National Medical Research Center of Oncology N.A. N.N. Petrov ( Site 0904), Saint Petersburg, Sankt-Peterburg
  - Republican Clinical Oncology Dispensary of Tatarstan MoH ( Site 0910), Kazan', Tatarstan, Respublika
- South Korea (4):
  - Chungbuk National University Hospital ( Site 1003), Cheongju-si, Chungcheongbuk-do [Chungbuk]
  - National Cancer Center ( Site 1002), Goyang-si, Kyonggi-do
  - Samsung Medical Center ( Site 1001), Seoul, Seoul-teukbyeolsi [Seoul]
  - Ulsan University Hospital ( Site 1000), Ulsan, Ulsan-Kwangyokshi
- Spain (5):
  - Hospital Universitari Vall d Hebron ( Site 1101), Barcelona, Barcelona [Barcelona]
  - Hospital Clinic de Barcelona ( Site 1100), Barcelona, Barcelona [Barcelona]
  - Hospital Son Llatzer ( Site 1105), Palma de Mallorca, Illes Balears [Islas Baleares]
  - Clinica Universitaria de Navarra ( Site 1102), Madrid
  - Hospital Universitario Virgen Macarena ( Site 1103), Seville
- United Kingdom (6):
  - Southampton General Hospital ( Site 1204), Southampton, Hampshire
  - Royal Free NHS Foundation Trust ( Site 1200), London, London, City of
  - Charing Cross Hospital ( Site 1208), London, London, City of
  - Beacon Centre ( Site 1203), Taunton, Somerset
  - Queen's Hospital ( Site 1201), Rom Valley, United Kingdom
  - Leeds Teaching Hospitals NHS Trust ( Site 1209), Leeds

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Jabbour SK, Lee KH, Frost N, Breder V, Kowalski DM, Pollock T, Levchenko E, Reguart N, Martinez-Marti A, Houghton B, Paoli JB, Safina S, Park K, Komiya T, Sanford A, Boolell V, Liu H, Samkari A, Keller SM, Reck M. Pembrolizumab Plus Concurrent Chemoradiation Therapy in Patients With Unresectable, Locally Advanced, Stage III Non-Small Cell Lung Cancer: The Phase 2 KEYNOTE-799 Nonrandomized Trial. JAMA Oncol. 2021 Jun 4;7(9):1-9. doi: 10.1001/jamaoncol.2021.2301. Online ahead of print. PMID 34086039
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with unresectable, locally advanced, Stage III non-small cell lung cancer (NSCLC), who had received no prior anticancer therapy for their disease were recruited into two cohorts.
Pre-assignment Details: Of 216 participants enrolled/allocated in the trial, 214 received treatment.
Groups:
- Pembrolizumab + cCRT + Paclitaxel + Carboplatin: Participants received 1 cycle of carboplatin area under the curve (AUC) 6 mg/mL/min with paclitaxel 200 mg/m^2 and pembrolizumab 200 mg on Day 1. Approximately 3 weeks later, participants received carboplatin AUC 2 mg/mL/min with paclitaxel 45 mg/ m^2 administered weekly for 6 weeks along with 2 cycles of pembrolizumab 200 mg administered every 3 weeks (Q3W) in conjunction with standard thoracic radiotherapy (TRT) (60 Gray [Gy] in 2 Gy fractions administered 5 days per week for 6 weeks). Participants then received 14 additional cycles of pembrolizumab 200 mg administered Q3W. 1 cycle=21 days.
- Pembrolizumab + cCRT + Pemetrexed + Cisplatin: Participants received 3 cycles of cisplatin 75 mg/m^2 with pemetrexed 500 mg/m^2 and pembrolizumab 200 mg on Day 1 of each cycle. Treatment was given in conjunction with standard TRT (60 Gy in 2 Gy fractions administered 5 days per week for 6 weeks) in cycles 2 and 3. Participants then received 14 additional cycles of pembrolizumab 200 mg administered Q3W. 1 cycle=21 days.
Period: Overall Study
Arm/Group | Pembrolizumab + cCRT + Paclitaxel + Carboplatin | Pembrolizumab + cCRT + Pemetrexed + Cisplatin
Started | 112 | 104
Treated | 112 | 102
Completed | 0 | 0
Not Completed | 112 | 104
Not completed — Participants Ongoing | 1 | 0
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Sponsor's Decision | 36 | 52
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 71 | 49

BASELINE CHARACTERISTICS:
Population: The analysis population consisted of all allocated participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab + cCRT + Paclitaxel + Carboplatin | Pembrolizumab + cCRT + Pemetrexed + Cisplatin | Total
Number analyzed (Participants) | 112 | 104 | 216
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.7 (9.1) | 63.2 (9.4) | 64.5 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 40 | 76
  Male | 76 | 64 | 140
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 101 | 84 | 185
  Unknown or Not Reported | 9 | 17 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 14 | 11 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 89 | 75 | 164
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 14 | 21

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Developed Grade 3 or Higher Pneumonitis
Description: Pneumonitis included the MedDRA preferred terms for radiation pneumonitis are acute interstitial pneumonitis, autoimmune lung disease, interstitial lung disease, pneumonitis, idiopathic pneumonia syndrome, organizing pneumonia, and immune-mediated pneumonitis. As per common terminology criteria for Adverse Events, version 4.0, pneumonitis was graded as follows: Grade (Gr) 1- asymptomatic, clinical or diagnostic observations only; intervention not indicated; Gr 2- symptomatic, medical intervention indicated, limiting instrumental activities of daily living (ADL); Gr 3- severe symptoms; limiting self-care activities of daily living (ADL), oxygen indicated; Gr 4- life-threatening respiratory compromise; urgent intervention indicated (e.g., tracheotomy or intubation); Gr 5- death.
Time Frame: Up to approximately 3 years
Population: The analysis population consisted of all participants who received at least one dose of study drug.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + cCRT + Paclitaxel + Carboplatin | Pembrolizumab + cCRT + Pemetrexed + Cisplatin
Number analyzed (Participants) | 112 | 102
Percentage of Participants | 8.0 [4.3 to 13.6] | 6.9 [3.3 to 12.5]

2. Primary Outcome: Overall Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: ORR was defined as the percentage of participants who experienced a complete response (CR; disappearance of all target lesions) or a partial response (PR; at least a 30% decrease in the sum of diameters of target lesions) and was assessed using modified RECIST 1.1 by blinded independent central review (BICR).
Time Frame: Up to approximately 3 years
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + cCRT + Paclitaxel + Carboplatin | Pembrolizumab + cCRT + Pemetrexed + Cisplatin
Number analyzed (Participants) | 112 | 102
Percentage of Participants | 71.4 [62.1 to 79.6] | 75.5 [66.0 to 83.5]

3. Secondary Outcome: Progression Free Survival (PFS) Per Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: PFS was defined as the time from the first dose of study treatment to the date of the first documentation of disease progression, as determined by BICR per RECIST 1.1 or death due to any cause (whichever occurred first). Disease progression was defined as at least 20 percent (%) increase (including an absolute increase of at least 5 millimeters [mm]) in the sum of diameter of target lesions, taking as reference the smallest sum, and/or unequivocal progression of existing non-target lesions, and/or appearance of 1 or more new lesions. PFS was estimated and analyzed using the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 5 1/2 years
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + cCRT + Paclitaxel + Carboplatin | Pembrolizumab + cCRT + Pemetrexed + Cisplatin
Number analyzed (Participants) | 112 | 102
Months | 29.0 [16.6 to 48.5] | 45.3 [17.9 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event.

4. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from enrollment to death due to any cause. OS was estimated and analyzed using the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 5 1/2 years
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + cCRT + Paclitaxel + Carboplatin | Pembrolizumab + cCRT + Pemetrexed + Cisplatin
Number analyzed (Participants) | 112 | 102
Months | 35.6 [26.1 to 44.2] | 56.7 [41.1 to NA] — NA= Upper limit not reached at time of data cut-off due to insufficient number of participants with an event.

5. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants with at least one AE was assessed.
Time Frame: Up to approximately 1 1/2 years
Population: The analysis population consisted of all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + cCRT + Paclitaxel + Carboplatin | Pembrolizumab + cCRT + Pemetrexed + Cisplatin
Number analyzed (Participants) | 112 | 102
Participants | 108 | 101

6. Secondary Outcome: Number of Participants Who Discontinued From Study Treatment Due to an AE
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinued treatment due to an AE was assessed.
Time Frame: Up to approximately 1 year
Population: The analysis population consisted of all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + cCRT + Paclitaxel + Carboplatin | Pembrolizumab + cCRT + Pemetrexed + Cisplatin
Number analyzed (Participants) | 112 | 102
Participants | 48 | 26

ADVERSE EVENTS:
Time Frame: For adverse events: Up to ~ 1 1/2 years. All-cause mortality (ACM): Up to ~ 5 1/2 years
Description: All-cause mortality includes all enrolled participants. AEs include participants who received ≥1 dose of study treatment. Per protocol, disease progression was not considered an AE, unless related to study treatment. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study treatment were excluded as AEs.
Arm/Group | Pembrolizumab + cCRT + Paclitaxel + Carboplatin | Pembrolizumab + cCRT + Pemetrexed + Cisplatin
All-Cause Mortality (participants affected / at risk) | 72/112 | 49/104
Serious Adverse Events (participants affected / at risk) | 66/112 | 46/102
Other Adverse Events (participants affected / at risk) | 106/112 | 100/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + cCRT + Paclitaxel + Carboplatin (N=112) | Pembrolizumab + cCRT + Pemetrexed + Cisplatin (N=102)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
Haematotoxicity (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypophysitis (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 2 (2) | 2 (2)
Death (General disorders) | 1 (1) | 0 (0)
Device related thrombosis (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 7 (9)
Sudden death (General disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatobiliary disease (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 2 (2) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Encephalitis (Infections and infestations) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 2 (3) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 14 (15) | 9 (11)
Pneumonia necrotising (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 4 (5) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertrophic osteoarthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Prerenal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (5)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + cCRT + Paclitaxel + Carboplatin (N=112) | Pembrolizumab + cCRT + Pemetrexed + Cisplatin (N=102)
Anaemia (Blood and lymphatic system disorders) | 44 (53) | 33 (40)
Leukopenia (Blood and lymphatic system disorders) | 15 (29) | 8 (11)
Lymphopenia (Blood and lymphatic system disorders) | 11 (13) | 12 (16)
Neutropenia (Blood and lymphatic system disorders) | 32 (50) | 23 (29)
Thrombocytopenia (Blood and lymphatic system disorders) | 17 (22) | 3 (3)
Tachycardia (Cardiac disorders) | 8 (9) | 3 (3)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 11 (13)
Vertigo (Ear and labyrinth disorders) | 6 (6) | 3 (3)
Hyperthyroidism (Endocrine disorders) | 9 (9) | 8 (9)
Hypothyroidism (Endocrine disorders) | 18 (19) | 15 (16)
Abdominal pain (Gastrointestinal disorders) | 8 (8) | 6 (7)
Abdominal pain upper (Gastrointestinal disorders) | 3 (4) | 7 (7)
Constipation (Gastrointestinal disorders) | 24 (28) | 27 (32)
Diarrhoea (Gastrointestinal disorders) | 27 (37) | 22 (27)
Dyspepsia (Gastrointestinal disorders) | 15 (17) | 7 (9)
Dysphagia (Gastrointestinal disorders) | 27 (31) | 16 (16)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (5) | 6 (6)
Nausea (Gastrointestinal disorders) | 28 (36) | 53 (77)
Odynophagia (Gastrointestinal disorders) | 11 (14) | 5 (5)
Oesophagitis (Gastrointestinal disorders) | 17 (20) | 24 (25)
Stomatitis (Gastrointestinal disorders) | 7 (8) | 6 (7)
Vomiting (Gastrointestinal disorders) | 10 (11) | 20 (23)
Asthenia (General disorders) | 20 (26) | 41 (60)
Chest pain (General disorders) | 7 (7) | 10 (12)
Chills (General disorders) | 6 (6) | 3 (3)
Fatigue (General disorders) | 39 (49) | 33 (38)
Mucosal inflammation (General disorders) | 6 (6) | 10 (10)
Pyrexia (General disorders) | 22 (30) | 13 (14)
Pneumonia (Infections and infestations) | 12 (14) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 8 (9) | 5 (5)
Urinary tract infection (Infections and infestations) | 7 (8) | 2 (2)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 13 (13) | 14 (15)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 18 (18) | 12 (12)
Radiation skin injury (Injury, poisoning and procedural complications) | 5 (5) | 8 (8)
Alanine aminotransferase increased (Investigations) | 8 (9) | 8 (9)
Aspartate aminotransferase increased (Investigations) | 8 (8) | 4 (6)
Blood creatinine increased (Investigations) | 6 (7) | 13 (17)
Blood urea increased (Investigations) | 3 (3) | 7 (9)
Lymphocyte count decreased (Investigations) | 11 (16) | 8 (12)
Neutrophil count decreased (Investigations) | 19 (23) | 13 (15)
Platelet count decreased (Investigations) | 16 (18) | 9 (15)
Weight decreased (Investigations) | 16 (16) | 14 (14)
White blood cell count decreased (Investigations) | 11 (17) | 11 (19)
Decreased appetite (Metabolism and nutrition disorders) | 24 (29) | 30 (34)
Dehydration (Metabolism and nutrition disorders) | 5 (6) | 6 (7)
Hyperglycaemia (Metabolism and nutrition disorders) | 9 (13) | 6 (11)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6 (8) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 9 (10) | 6 (8)
Hyponatraemia (Metabolism and nutrition disorders) | 10 (15) | 3 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 (22) | 11 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (8) | 5 (7)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6 (8) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (14) | 8 (9)
Dizziness (Nervous system disorders) | 9 (11) | 9 (11)
Dysgeusia (Nervous system disorders) | 10 (11) | 8 (8)
Headache (Nervous system disorders) | 9 (9) | 13 (18)
Neuropathy peripheral (Nervous system disorders) | 15 (15) | 5 (5)
Paraesthesia (Nervous system disorders) | 6 (7) | 4 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 12 (13) | 1 (1)
Insomnia (Psychiatric disorders) | 18 (21) | 7 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 31 (36) | 29 (37)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24 (28) | 18 (19)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 8 (8)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 16 (19) | 17 (19)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 9 (9)
Alopecia (Skin and subcutaneous tissue disorders) | 35 (35) | 6 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 15 (19) | 16 (18)
Rash (Skin and subcutaneous tissue disorders) | 22 (27) | 14 (16)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (2)
Hypertension (Vascular disorders) | 6 (6) | 5 (7)
Hypotension (Vascular disorders) | 11 (11) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-05): https://cdn.clinicaltrials.gov/large-docs/84/NCT03631784/Prot_SAP_001.pdf